CLINICAL TRIAL: NCT06916507
Title: German Real-World Evidence Study on the Effectiveness of Foslevodopa/Foscarbidopa at Initial Stages of Advanced Parkinson's Disease: Motor Symptoms, Quality of Life, Psychosocial Functioning and Work Ability
Brief Title: Study to Assess Real Life Effectiveness of Foslevodopa/Foscarbidopa in Adult German Participants at Initial Stages of Advanced Parkinson's Disease (EARLY-FOS)
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P25-278
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Foscarbidopa/Foslevodopa
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Foslevodopa/Foscarbidopa: Participants will receive Foslevodopa/Foscarbidopa as prescribed by their physician according to local label.

SUMMARY:
Parkinson's disease (PD) is a neurological condition, which affects the brain. PD gets worse over time, but how quickly it progresses varies a lot from person to person. Some symptoms of PD are tremors, stiffness, and slowness of movement. This study will assess how effective foscarbidopa/ foslevodopa is in treating German adult participants at initial stages of advanced Parkinson's disease under routine clinical practice.

Foslevodopa/Foscarbidopa is an approved drug for the treatment of Parkinson's Disease. Approximately 125 adult participants who are prescribed Foslevodopa/Foscarbidopa by their doctors will be enrolled across approximately 20 sites in Germany.

Participants will receive Foslevodopa/Foscarbidopa subcutaneous infusion as prescribed by their physician. Participants will be followed for up to 12 months.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of levodopa-responsive idiopathic Parkinson's disease
* Eligibility for foscarbidopa/foslevodopa (LDp/CDp) therapy in accordance with the approved local label
* Participant must be an adult male or female, 18-64 years of age
* Time since beginning of motor fluctuations ≤ 3 years
* The Hoehn and Yahr (H&Y) stage < 3 in the on-medication condition
* Decision to treat with LDp/CDp made by the clinician prior to any decision to approach the participant to participate in this study

Exclusion Criteria:

* Previous Exposure to any device-aided therapy (DAT).
* Any condition included in the contraindications section of the approved local LDp/CDp label.
* Participants with Mini mental state examination (MMSE) score < 24

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants with advanced Parkinson's disease with time since the beginning of motor fluctuations ≤3 years and the Hoehn and Yahr (H&Y) stage < 3 in the on-medication condition treated with foslevodopa/foscarbidopa according to label in Germany
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in OFF Time (hours) | Up To 12 months
  The mean change from baseline to each scheduled visit in the number of hours spent in OFF time will be estimated using a mixed-effect model repeated-measures (MMRM).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (13):
- Germany (13):
  - Universitaetsklinikum Heidelberg /ID# 274164, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen /ID# 275828, Tübingen, Baden-Wurttemberg
  - Praxis Prof. Kassubek/Prof. Riecker /ID# 274165, Ulm, Baden-Wurttemberg
  - Parkinson-Klinik Ortenau GmbH&Co KG /ID# 274161, Wolfach, Baden-Wurttemberg
  - Klinikum der Universitaet Muenchen Grosshadern /ID# 274168, Munich, Bavaria
  - Klinikum Ernst von Bergmann /ID# 274176, Potsdam, Brandenburg
  - Universitaetskliniken Giessen und Marburg /ID# 274224, Marburg, Hesse
  - Knappschaftskrankenhaus Bottrop /ID# 274284, Bottrop, North Rhine-Westphalia
  - Cellitinnen-NTC Neurologisches Therapiecentrum /ID# 277865, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 274167, Dresden, Saxony
  - Krankenhaus Martha-Maria Halle-Dölau /ID# 274174, Halle, Saxony-Anhalt
  - Praxis MD Oehlwein /ID# 274222, Gera, Thuringia
  - Asklepios Fachklinikum Stadtroda /ID# 274162, Stadtroda, Thuringia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P25-278